CLINICAL TRIAL: NCT03167138
Title: Treatment of Chronic Shoulder Pain in Persons With Spinal Cord Injury Using Injection With Autologous Micro-Fragmented Adipose Tissue Under Ultrasound Guidance
Brief Title: Micro-Fragmented Adipose Tissue (Lipogems®) Injection for Chronic Shoulder Pain in Persons With Spinal Cord Injury
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Kessler Foundation (Other)
Responsible Party: Principal Investigator, Trevor Dyson-Hudson, M.D., Director, Spinal Cord Injury Research, Kessler Foundation
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R-957-17
Record Dates: First submitted 2017-05-24; First posted 2017-05-25 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Shoulder Pain; Shoulder Impingement Syndrome; Rotator Cuff Impingement Syndrome; Rotator Cuff Tendinitis; Rotator Cuff Syndrome of Shoulder and Allied Disorders; Spinal Cord Injuries
Keywords: Shoulder pain; Rotator cuff disease; Spinal cord injuries; Mesenchymal stromal cells; Regenerative medicine; Rehabilitation
MeSH Terms: conditions — Shoulder Pain; Shoulder Impingement Syndrome; Rotator Cuff Injuries; Spinal Cord Injuries

STUDY DESIGN:
Intervention Model Description: Single Group Assignment
Masking Description: No masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Autologous micro-fragmented adipose tissue (Experimental): Injection (under ultrasound guidance) of autologous micro-fragmented adipose tissue obtained from abdominal region or thighs using the Lipogems® system.
  Interventions: Biological: Autologous micro-fragmented adipose tissue; Device: Lipogems system

INTERVENTIONS:
Biological: Autologous micro-fragmented adipose tissue — Micro-fragmented adipose tissue is obtained from abdominal region or thighs using the Lipogems® system and injected into the injury site under ultrasound guidance.
  Other Names: Lipogems
Device: Lipogems system — The Lipogems® system is a non-enzymatic method to obtain micro-fragmented adipose tissue from the abdominal region or thighs for injection into the injury site.
  Other Names: Lipogems technological process

SUMMARY:
Rotator cuff disease (i.e., rotator cuff tendinopathy or tear) is a common cause of shoulder pain in persons with chronic spinal cord injury (SCI). It usually resolves with non-operative treatments such as pharmacological agents and physical therapy; however, when this fails, rotator cuff surgery may be the only option. Autologous adipose tissue injection has recently emerged as a promising new treatment for joint pain and soft tissue injury. Adipose can be used to provide cushioning and filling of structural defects and has been shown to have an abundance of bioactive elements and regenerative perivascular cells (pericytes). The purpose of this study is to explore the safety and efficacy of autologous, micro-fragmented adipose tissue (Lipogems®) injection under ultrasound guidance for chronic shoulder pain in persons with SCI.

DETAILED DESCRIPTION:
This is an exploratory pilot study to determine the safety and efficacy of autologous, micro-fragmented adipose tissue (Lipogems®) injection under ultrasound guidance for chronic, nonresponsive shoulder pain due to rotator cuff disease (i.e., rotator cuff tendinopathy) in persons with spinal cord injury (SCI). Twelve (12) persons with SCI who have chronic shoulder pain for longer than 6 months in spite of completing conservative treatment who are diagnosed with rotator cuff disease on examination. Micro-fragmented adipose tissue will be obtained by using a minimal manipulation technique in a closed system (Lipogems®), without the addition of enzymes or any additives. The final product will consist of micronized fat tissue yielding fat clusters with preserved vascular stroma of about 500 microns with intact stromal vascular niches and harboring regenerative cellular elements. Approximately 6 mL of micro-fragmented adipose will be injected into the tendon with a 22-gauge needle under continuous ultrasound guidance. No other biological or pharmacological agents will be used in combination with the micro-fragmented adipose. After 24 hours, subjects will be given a standardized stretching protocol to follow for 4 weeks followed by a formal strengthening program. Participants will be followed for adverse events and changes in shoulder pain intensity on an 11-point numerical rating scale (NRS; 0-10, with anchors "no pain" and "pain as bad as you can imagine"); the Wheelchair User's Shoulder Pain Index (WUSPI; 15-item disease-specific functional measure of shoulder pain in persons with SCI); the Brief Pain Inventory interference items (BPI-I7; a subscale of 7 items measuring interference with general activity, sleep, mood, relationships, etc.); and a 5-point subject global impression of change (SGIC) scale. Subjects will be examined at 1 month, 2 months, 3 months, and 6 months after the treatment. Follow-up shoulder ultrasound will be performed at 6 months.

ELIGIBILITY:
Inclusion Criteria:

* The subject is male or female, 18 to 60 years of age, inclusive.
* The subject has neurological impairment secondary to a spinal cord injury that occurred at least twelve (12) months prior to the Screening Visit and the level of the injury is between C5 and L5, inclusive.
* The subject is non-ambulatory except for exercise purposes and uses a manual or power wheelchair as his/her primary means of mobility (> 40 hours/week).
* The subject currently has chronic shoulder pain due to rotator cuff disease in spite of at least 6 months of conservative treatment (Note: rotator cuff disease will be defined as pain over the anterior shoulder, with direct palpation and pain at the shoulder with provocative tests for rotator cuff disease that is confirmed by tendinopathic changes on ultrasound imaging).
* The average shoulder pain intensity during the week leading up to the Screening Visit should be at least 4 out of 10 on an 11-point numerical rating scale (NRS; 0, no pain; 10, maximum pain imaginable).
* The subject is able and willing to comply with the protocol.
* The subject is able to and has voluntarily given informed consent prior to the performance of any study-specific procedures.

Exclusion Criteria:

* The subject reports prior Lipogems treatment in the same shoulder.
* The subject reports a history of systemic disorders, such as diabetes or rheumatoid arthritis.
* The subject has contra-indications to the procedure, such as infection, coagulopathy, or is currently taking anti-coagulants.
* The subject reports having a glucocorticoid injection in the past 4 weeks.
* The subject is pregnant (documented by a urine pregnancy test).
* The subject has any medical condition, including psychiatric disease, which would interfere with the interpretation of the study results or the conduct of the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-07-14 (Actual); Primary Completion 2019-09-06 (Actual); Study Completion 2020-02-21 (Estimated)

PRIMARY OUTCOMES:
Numerical Rating Scale | Baseline and 4 weeks, 8 weeks, 12 weeks, and 24 weeks after the treatment.
  Shoulder pain intensity will also be assessed weekly using a numerical rating scale (NRS). Subjects will be asked to rate their average pain, most severe pain, and least severe pain during the past week using an 11-point scale (i.e. 0-10) anchored at the ends by "no pain" and "pain as bad as you can imagine." An 11-point NRS measure of pain intensity allows for comparison across clinical trials of chronic pain treatment and is recommended as a core outcome measure for chronic pain clinical trials.

SECONDARY OUTCOMES:
Wheelchair User's Shoulder Pain Index (WUSPI) | Baseline and 4 weeks, 8 weeks, 12 weeks, and 24 weeks after the treatment.
  The WUSPI is a 15-item self-report instrument that measures shoulder pain intensity in wheelchair users during various ADLs, such as transfers, loading a wheelchair into a car, wheelchair mobility, dressing, bathing, overhead lifting, driving, performing household chores, and sleeping. Each item is scored using a 10cm visual analog scale (VAS) which is anchored at the ends with "no pain" and "worst pain ever experienced." Individual item scores are summed to arrive at a total index score, which ranges from 0 to 150.
Patient Global Impression of Change | Baseline and 4 weeks, 8 weeks, 12 weeks, and 24 weeks after the treatment.
  Subjects will be asked to rate on a 7-point scale overall impression following treatment as compared to the previous measurement interval. The 7-point PGIC scale (anchored by "very much improved" and "very much worse") is used to measure global treatment effect.
Brief Pain Inventory interference items (BPI-I7) | Baseline and 4 weeks, 8 weeks, 12 weeks, and 24 weeks after the treatment.
  The Brief Pain Inventory (BPI) was developed by Cleeland, and has been used in a number of investigations of chronic pain. Its pain interference subscale has been used in several investigations of pain in SCI. In its original version the subscale (BPI-I7) consisted of 7 items measuring interference with general activity, sleep, mood, relationships, etc.). For uses with an SCI sample, in item 3 of BPI-I7, ''walking ability'' is replaced by "ability to get around."
Physical Examination of the Shoulder Score (PESS) | Baseline and 4 weeks, 8 weeks, 12 weeks, and 24 weeks after the treatment.
  The Physical Examination of the Shoulder Score (PESS) is obtained by performing a series of eleven commonly used physical examination maneuvers for rotator cuff disease and shoulder pain that are graded 0 (no pain), 1 (equivocal for pain), or 2 (pain present).

CONTACTS AND LOCATIONS:
Overall Officials: Trevor A. Dyson-Hudson, M.D., Principal Investigator — Kessler Foundation
Locations (1):
- Kessler Institute for Rehabilitation, West Orange, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hogaboom N, Malanga G, Cherian C, Dyson-Hudson T. A pilot study to evaluate micro-fragmented adipose tissue injection under ultrasound guidance for the treatment of refractory rotator cuff disease in wheelchair users with spinal cord injury. J Spinal Cord Med. 2021 Nov;44(6):886-895. doi: 10.1080/10790268.2021.1903140. Epub 2021 Apr 8. PMID 33830898